CLINICAL TRIAL: NCT02032004
Title: Double-blind, Randomized, Sham-procedure-controlled, Parallel-Group Efficacy and Safety Study of Allogeneic Mesenchymal Precursor Cells (Rexlemestrocel-L) in Chronic Heart Failure Due to LV Systolic Dysfunction (Ischemic or Nonischemic) Dream HF-1
Brief Title: Efficacy and Safety of Allogeneic Mesenchymal Precursor Cells (Rexlemestrocel-L) for the Treatment of Heart Failure.
Acronym: DREAM HF-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mesoblast, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mesoblast, Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MSB-MPC-CHF001
Record Dates: First submitted 2014-01-08; First posted 2014-01-09 (Estimated); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: Chronic Heart Failure
Keywords: Chronic Heart Failure; CHF; Left Ventricular Systolic Dysfunction; Ischemic Heart Failure; Nonischemic Heart Failure; Stem Cells; Allogeneic Mesenchymal Precursor Cells
MeSH Terms: conditions — Ventricular Dysfunction, Left

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Allogeneic Mesenchymal Precursor Cells (Experimental): Participants randomly assigned to treatment will undergo a single index cardiac catheterization involving transendocardial delivery of rexlemestrocel-L into the myocardium at a cell injection center by an interventional cardiology team not involved with review or assessment of subsequent study results.
  Interventions: Biological: Allogeneic Mesenchymal Precursor Cells (MPCs)
- Control Treatment (Sham Comparator): Participants randomly assigned to control treatment will undergo a single cardiac catheterization involving a scripted sham cardiac mapping and cell delivery procedure at a cell injection center by an interventional cardiology team not involved with review or assessment of subsequent study results.
  Interventions: Other: Sham Comparator

INTERVENTIONS:
Biological: Allogeneic Mesenchymal Precursor Cells (MPCs) — Rexlemestrocel-L consists of human bone marrow-derived allogeneic MPCs isolated from bone mononuclear cells with anti-STRO-3 antibodies, expanded ex vivo, and cryopreserved
  Other Names: MPCs; rexlemestrocel-L
  Arms: Allogeneic Mesenchymal Precursor Cells
Other: Sham Comparator — The sham procedure will be staged to script and will not include actual cardiac mapping or delivery of rexlemestrocel-L.
  Arms: Control Treatment

SUMMARY:
The primary objective of this study is to determine whether transendocardial delivery of allogeneic human bone marrow-derived mesenchymal precursor cells (MPCs [rexlemestrocel-L]) is effective in the treatment of chronic heart failure (HF) due to left ventricular (LV) systolic dysfunction.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy and safety of a single transendocardial delivery in the cardiac catheterization laboratory of human bone marrow-derived allogeneic MPCs (rexlemestrocel-L) for improvement in clinical outcomes (heart failure major adverse cardiac events [HF-MACE]), preventing further adverse cardiac remodeling (left ventricular end systolic volume [LVESV] and left ventricular end-diastolic volume [LVEDV]), and increasing exercise capacity (six-minute walking test [6MWT]) in patients with chronic HF due to LV systolic dysfunction of either ischemic or nonischemic etiology who have received optimal medical/revascularization therapy.

ELIGIBILITY:
Inclusion Criteria:

* The patient is 18 to 80 years of age, inclusive; both men and women will be enrolled.
* The patient has a diagnosis of chronic HF of ischemic or nonischemic etiology for at least 6 months
* The patient is on stable, optimally tolerated dosages of HF therapies including beta-blockers (approved for country-specific usage), angiotensin-converting enzyme (ACE) inhibitors or angiotensin-receptor blockers (ARBs), and/or aldosterone antagonists, without change in dose for at least 1 month before study intervention
* The patient is on a stable, outpatient, oral diuretic dosing regimen in which the patient remains clinically stable during screening.
* Other Criteria apply, please contact the investigator

Exclusion Criteria:

* The patient has NYHA Functional Class I or Functional Class IV symptoms.
* Other Criteria apply, please contact the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 566 (Actual)
Dates: Start 2014-02-14 (Actual); Primary Completion 2020-05-29 (Actual); Study Completion 2020-05-29 (Actual)

PRIMARY OUTCOMES:
Time to recurrent non-fatal decompensated heart failure major adverse cardiac events (HF-MACE) that occur prior to the first terminal cardiac event (TCE). | 6 Month minimum

SECONDARY OUTCOMES:
Time-to-first terminal cardiac event (TCE) | 6 Month minimum
Time-to-hospital admissions for non-fatal decompensated HF events | 6 Month minimum
Time-to-urgent care outpatient HF visits | 6 Month minimum
Time-to-successfully resuscitated cardiac death (RCD) events | 6 Month minimum
Total length of in-hospital stay in intensive care unit for non-fatal decompensated HF events | 6 Month minimum
Time-to-first HF-MACE (composite of hospital admissions for decompensated HF, urgent care outpatient HF visit, and successfully RCD events) | 6 Month minimum
Time-to-first HF-MACE (composite of hospital admissions for decompensated HF, urgent care outpatient HF visit, successfully RCD events or TCE) | 6 Month minimum
Time-to-cardiac death | 6 Month minimum
Time-to-all-cause death | 6 Month minimum
Time-to-first non-fatal MI (myocardial infarction), non-fatal CVA (cerebrovascular attack) or coronary artery revascularization | 6 Month minimum
Left Ventricular (LV) remodeling in LVESV determined by 2-D echocardiography | Screening, day 0 (post-procedure), months 3, 6, and 12, and every 12 months thereafter during study conduct (6 Month minimum)
Correlations between baseline LVESV <=100 mL and LVESV >100 mL and clinical outcomes | 6 Month minimum
Correlations between baseline LVESV <=100 mL and LVESV >100 mL and change in Month 6 to baseline LVESV and clinical outcomes | 6 Month minimum
LV remodeling in LVEDV determined by 2-D echocardiography | Screening, day 0 (post-procedure), months 3, 6, and 12, and every 12 months thereafter during study conduct (6 Month minimum)
Overall Left Ventricular systolic performance as assessed by left ventricular ejection fraction (LVEF [radionuclide ventriculography {RVG} or echocardiogram]) | Screening, day 0 (post-procedure), months 3, 6, and 12, and every 12 months thereafter during study conduct (6 Month minimum)
Functional exercise capacity as assessed by 6 Minute Walk Test | Screening, months 3, 6, and 12, and every 12 months thereafter during study conduct (6 Month minimum)
Functional status by New York Heart Association (NYHA) class | Screening, months 3, 6, and 12, and every 12 months thereafter during study conduct (6 Month minimum)
Quality of Life Measure - Minnesota Living With Heart Failure (MLHF) questionnaire | Screening, months 3, 6, and 12, and every 6 months thereafter during study conduct (6 Month minimum)
Quality of Life Measure - European Quality of Life (EuroQoL) 5-dimensional (EQ-5D) questionnaire | Screening, months 3, 6, and 12, and every 6 months thereafter during study conduct (6 Month minimum)
Safety as assessed by occurrence of adverse events related to the index cardiac catheterization on Day 0 | Day 0 through discharge from Day 0 hospitalization
Safety as assessed by occurrence of treatment-emergent adverse events | Screening through 6 Month minimum
Safety as assessed by clinical laboratory tests (serum chemistry - ALT, AST, alkaline phosphate, GGT, LDH, BUN, creatinine, uric acid, total bilirubin - and hematology - hematocrit, hemoglobin, WBCs, eosinophils, ANC, platelet count) | Screening, day 0 (post-procedure), day 10, months 1, 3, 6, and 12, and every 6 months thereafter during study conduct (6 Month minimum)
  ALT (alanine transaminase), AST (aspartate aminotransferase), GGT (gamma-glutamyl transferase), LDH (lactate dehydrogenase), BUN (blood urea nitrogen), WBCs (white blood cells), ANC (absolute neutrophil count)
Safety as assessed by urinalysis (blood, glucose, ketones, total protein) | Screening, day 10, months 1, 3, 6, and 12, and every 6 months thereafter during study conduct (6 Month minimum)
Safety as assessed by vital signs (pulse, systolic blood pressure [BP], diastolic BP) | Screening, day 0 (pre and post-procedure), day 1, day 10, months 1, 3, 6, and 12, and every 6 months thereafter during study conduct (6 Month minimum)
Safety as assessed by 12-lead electrocardiogram (ECG) findings - QT interval with Fridericia's correction (QTcF), heart rate-corrected QT interval (QTcB), QT, Q wave, R wave and S wave (QRS) complex, HR and T waves. | Screening, day 0 (pre and post-procedure), day 1, day 10, months 1, 3, 6, and 12, and every 6 months thereafter during study conduct (6 Month minimum)
Safety as assessed by telemetry monitoring findings (clinically significant arrhythmias) | Day 0 through Day 0 overnight post-procedure
Safety as assessed by rhythm analysis (specifically, ventricular arrhythmias) by interrogation of any implanted device capable of defibrillation | Day 10, months 1, 3, 6, and 12, and every 6 months thereafter during study conduct (6 Month minimum)
Safety as assessed by 24-hr Holter monitoring (HR, rate & duration of arrhythmias, a-fib average rate, supra- & ventricular ectopy singles/couplets/runs/totals, sustained & non-sustained ventricular tachycardia, longest pauses RR duration, total pauses) | Screening, day 0 (post-procedure), day 10, months 1 and 3
Safety as assessed by physical examination findings judged as clinically significant changes from baseline by the investigator or newly occurring abnormalities (including weight) | Screening, month 12 and every 12 months thereafter until study conclusion (weight measured at screening, day 0 - pre and post-procedure, day 1, day 10, months 1, 3, 6 and 12 and every 6 months thereafter)
Safety as assessed by important cardiovascular events from adjudicated data | 6 Month minimum

OTHER OUTCOMES:
Pharmacodynamics Measures (N-terminal (NT)-pro hormone BNP [NT-proBNP] and high-sensitivity C-reactive protein [hs-CRP]) | Screening, months 3, 6, 12 and every 12 months thereafter until study conclusion
Pharmacogenomics (PGx) Analysis | Screening (only from those subjects who provide consent to participate in PGx sample collection)
Immunogenicity Measures (panel reactive antibodies, donor specific antibody, if panel-reactive antibody (PRA) test is positive, antibodies against bovine and murine products) | Screening, day 10, months 1, 3, 6, and 12

CONTACTS AND LOCATIONS:
Overall Officials: Fred Grossman, DO, Study Director — Mesoblast, Ltd.
Locations (59):
- United States (56):
  - Mesoblast Investigational Site 10757 - Cardiology, P.C., Birmingham, Alabama
  - Mesoblast Investigational Site 13262 - University of Alabama at Birmingham Hospital, Birmingham, Alabama
  - Mesoblast Investigational Site 10779 - Mercy Gilbert Medical Center, Gilbert, Arizona
  - Mesoblast Investigational Site 10786 - Cardiovascular Associates of Mesa, Mesa, Arizona
  - Mesoblast Investigational Site 10756 - Mayo Clinic, Phoenix, Arizona
  - Mesoblast Investigational Site 13023 - University of Arizona Medical Center, Tucson, Arizona
  - Mesoblast Investigational Site 10754 - University of California, San Diego, La Jolla, California
  - Mesoblast Investigational Site 10759 - Scripps Clinic, La Jolla, California
  - Mesoblast Investigational Site 13265 - University of California, Los Angeles, Los Angeles, California
  - Mesoblast Investigational Site 10775 - Cedars-Sinai Medical Care Foundation, Los Angeles, California
  - Mesoblast Investigational Site 10778 - Orange County Cardiology, Orange, California
  - Mesoblast Investigational Site 13031 - St. John's Regional Medical Center, Oxnard, California
  - Mesoblast Investigational Site 13275 - Stanford University Hospital, Stanford, California
  - Mesoblast Investigational Site 13267 - Bethesda Heart Hospital, Boynton Beach, Florida
  - Mesoblast Investigational Site 10780 - Morton Plant Hospital, Clearwater, Florida
  - Mesoblast Investigational Site 10760 - Shands Hospital, University of Florida, Gainesville, Florida
  - Mesoblast Investigational Site 13273 - University of Florida Health, Jacksonville, Florida
  - Mesoblast Investigational Site 10768 - University of Miami, Miami, Florida
  - Mesoblast Investigational Site 13280, Orlando, Florida
  - Mesoblast Investigational Site 13264 - Florida Hospital Pepin Heart Institute, Tampa, Florida
  - Mesoblast Investigational Site 13027 - Emory University School of Medicine, Atlanta, Georgia
  - Mesoblast Investigational Site 10765 - Georgia Regents University, Augusta, Georgia
  - Mesoblast Investigational Site 10772 - University Cardiologist, Rush University Medical Center, Chicago, Illinois
  - Mesoblast Investigational Site 13030 - University of Iowa, Iowa City, Iowa
  - Mesoblast Investigational Site 10783 - Gill Heart Institute, University of Kentucky, Lexington, Kentucky
  - Mesoblast Investigational Site 13022 - University of Louisville, Louisville, Kentucky
  - Mesoblast Investigational Site 13266, New Orleans, Louisiana
  - Mesoblast Investigational Site 10782, Boston, Massachusetts
  - Mesoblast Investigational Site 10766 - Michigan Cardiovascular Institute, Saginaw, Michigan
  - Mesoblast Investigational Site 10762 - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Mesoblast Investigational Site 10761 - Mayo Clinic, Rochester, Minnesota
  - Mesoblast Investigational Site 13281, Las Vegas, Nevada
  - Mesoblast Investigational Site 13263 - RWJ Barnabas Heart Center, Newark, New Jersey
  - Mesoblast Investigational Site 10776 - Columbia University Medical Center, New York, New York
  - Mesoblast Investigational Site 13026 - Sanger Heart and Vascular Institute, Carolinas Healthcare System, Charlotte, North Carolina
  - Mesoblast Investigational Site 10781 - Duke University, Durham, North Carolina
  - Mesoblast Investigational Site 10758 - The Christ Hospital, Cincinnati, Ohio
  - Mesoblast Investigational Site 10770 - University of Cincinnati, Cincinnati, Ohio
  - Mesoblast Investigational Site 10773, Cleveland, Ohio
  - Mesoblast Investigational Site 13278 - OhioHealth Research Institute, Columbus, Ohio
  - Mesoblast Investigational Site 10785 - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Mesoblast Investigational Site 13261 - University of Pennsylvania, Philadelphia, Pennsylvania
  - Mesoblast Investigational Site 10767 - Temple University Hospital, Philadelphia, Pennsylvania
  - Mesoblast Investigational Site 13277, Philadelphia, Pennsylvania
  - Mesoblast Investigational Site 10774 - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Mesoblast Investigational Site 10777 - Stern Cardiovascular Foundation, Germantown, Tennessee
  - Mesoblast Investigational Site 13024 - Austin Heart, PLLC, Austin, Texas
  - Mesoblast Investigational Site 13274 - Soltero CV Research Center, Baylor Scott & White Research Institute, Dallas, Texas
  - Mesoblast Investigational Site 10755 - Texas Heart Institute, Houston, Texas
  - Mesoblast Investigational Site 13268 - Houston Methodist Hospital, Houston, Texas
  - Mesoblast Investigational Site 10763 - University Hospital, Salt Lake City, Utah
  - Mesoblast Investigational Site 10771 - Heart & Vascular Research, Swedish Medical Center, Seattle, Washington
  - Mesoblast Investigational Site 10764 - University of Wisconsin, Madison, Wisconsin
  - Mesoblast Investigational Site 10769 - Aurora Healthcare, Milwaukee, Wisconsin
  - Mesoblast Investigational Site 13279, Milwaukee, Wisconsin
  - Mesoblast Investigational Site 10789 - Aspirus Research Institute, Wausau, Wisconsin
- Canada (3):
  - Mesoblast Investigational Site 11027, Edmonton, Alberta
  - Mesoblast Investigational Site 11024 - Victoria Heart Institute Foundation, Victoria, British Columbia
  - Mesoblast Investigational Site 11025 - St. Michael's Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Borow KM, Yaroshinsky A, Greenberg B, Perin EC. Phase 3 DREAM-HF Trial of Mesenchymal Precursor Cells in Chronic Heart Failure. Circ Res. 2019 Jul 19;125(3):265-281. doi: 10.1161/CIRCRESAHA.119.314951. Epub 2019 Jul 18. PMID 31318648